CLINICAL TRIAL: NCT03583086
Title: Phase 1/2 Study to Evaluate the Safety and Preliminary Activity of Nivolumab in Combination With Vorolanib in Patients With Refractory Thoracic Tumors
Brief Title: Phase I/II Eval Safety & Prelim Activity Nivolumab Comb W/Vorolanib Pts W/Refractory Thoracic Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Xcovery Holdings, Inc. (Industry)
Responsible Party: Principal Investigator, Kathryn Beckermann, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 1802; CA209-982 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Thymic Carcinoma; Non-small Cell Lung Cancer; Refractory Thoracic Tumors; Small-Cell Lung Cancer
MeSH Terms: conditions — Thymoma; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — vorolanib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Escalation (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab
- Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab
- Dose Expansion - Non Small-Cell-Lung Cancer Naive (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab
- Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab
- Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab
- Dose Expansion - Thymic Carcinoma (Experimental): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Interventions: Drug: Vorolanib; Biological: Nivolumab

INTERVENTIONS:
Drug: Vorolanib — Given by mouth
Biological: Nivolumab — Given by IV

SUMMARY:
This is a two-agent, open-label, non-randomized, Phase 1/2 dose escalation and dose expansion study of combinatorial oral vorolanib plus infusional nivolumab in patients with Non-Small Cell Lung Cancer naïve to checkpoint inhibitor therapy, Non-Small Cell Lung Cancer who have progressed on checkpoint inhibitor therapy, Small Cell Lung Cancer ( who have progressed on platinum-based chemotherapy, and thymic carcinoma.

DETAILED DESCRIPTION:
Primary Objectives:

* Phase I: To assess the safety and tolerability of nivolumab and vorolanib in combination in patients with refractory non small cell lung cancer naïve to checkpoint inhibitor therapy, non small cell lung cancer progressed on prior checkpoint inhibitor therapy considered primary refractory, non small cell lung cancer progressed on prior checkpoint inhibitor therapy considered acquired resistance, small cell lung cancer progressed on platinum-based chemotherapy, and thymic carcinoma.
* Phase II: To evaluate the efficacy as measured by response to the combination nivolumab and vorolanib in patients with refractory non small cell lung cancer naïve to checkpoint inhibitor therapy, non small cell lung cancer progressed on prior checkpoint inhibitor therapy considered primary refractory, non small cell lung cancer progressed on prior checkpoint inhibitor therapy considered acquired resistance, small cell lung cancer progressed on platinum-based chemotherapy, and thymic carcinoma as compared to historical controls.

Secondary Objectives:

* Phase I: To assess antitumor activity as measured by response rate for this novel combination.
* Phase II: To assess, safety, progression free survival and overall survival

Exploratory Objectives:

• To assess the effects of combinatorial treatment on specific pharmacodynamic and pharmacogenetic biomarkers including PD-L1 expression and tumor mutation burden.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent.
* Male or female ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Having progressed on at least one prior line of therapy, or refused chemotherapy, histologically or cytologically confirmed diagnosis of one of the following:

Dose Escalation and Expansion Cohorts:

* Checkpoint Inhibitor Naïve Non-Small Cell Lung Cancer patients must have progressed on front-line cytotoxic chemotherapy or have refused chemotherapy and may have received up to three prior treatment regimens for stage IV disease provided no regimens included an anti-PD1 or PD-L1 agent or an oral VEGF TKI. Prior bevacizumab or ramucirumab is allowed.
* Progressed on Checkpoint Inhibitor Non-Small Cell Lung Cancer patients must have progressed on front-line or second checkpoint inhibitor therapy and may have received up to three prior treatment regimens for stage IV disease provided no regimens included an oral VEGF TKI. Prior bevacizumab or ramucirumab is allowed.
* Patients with EGFR, ALK, ROS1 and BRAF NSCLC must have progressed on an oral TKI and may have received an unlimited number of prior regimens.
* Thymic carcinoma patients must not be eligible for surgical resection at the time of enrollment and may have received any number of prior lines of therapy provided no regimens included an anti-PD1 or PD-L1 agent or an oral VEGF TKI. Prior bevacizumab or ramucirumab is allowed.
* Small Cell Lung Cancer patients must have progressed on platinum-based chemotherapy and may have received up to three prior lines of therapy for stage IV disease provided no prior regimen included an oral VEGF TKI; prior regimens can include an anti-PD-1 or PD-L1 agent.

  * At least one measureable lesion as defined by RECIST 1.1 which can be followed by CT or MRI.
  * Adequate organ function prior to first dose of protocol-indicated treatment, including:
* Absolute neutrophil count (ANC) ≥ 1,500/µL
* Platelets ≥ 100,000/µL
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine ≤ 1.5 times institutional upper limit of normal (ULN), or calculated creatinine clearance ≥ 40 mL/min (per the Cockcroft-Gault formula)
* Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 3.0 mg/dL)
* Alanine aminotransferase and aspartate aminotransferase ≤ 2.5 x ULN, (≤ 5.0 x ULN with documented liver metastases)

  * Women must not be breastfeeding.
  * Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to receiving first dose of protocol-indicated treatment.
* Women of childbearing potential is defined as any female who has experienced menarche who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal.
* Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological causes.
* If menopausal status is considered for the purpose of evaluating childbearing potential, women < 62 years of age must have a documented serum follicle stimulating hormone (FSH) level within laboratory reference range for postmenopausal women, in order to be considered postmenopausal and not of childbearing potential.

  * Women of childbearing potential must agree to follow instructions for acceptable contraception Appendix 5 from the time of signing consent, and for 23 weeks after their last dose of protocol-indicated treatment.
  * Men not azoospermic who are sexually active with women of childbearing potential must agree to follow instructions for acceptable contraception (Appendix 5), from the time of signing consent, and for 31 weeks after their last dose of protocol-indicated treatment.

Exclusion Criteria:

* ≤ 28 days before first dose of protocol-indicated treatment:

  * Anti-cancer treatment with bevacizumab.
  * Major surgery requiring general anesthesia or significant traumatic injury.
* ≤ 14 days before first dose of protocol-indicated treatment:

  * Anti-cancer therapy with an approved or investigational agent (including chemotherapy, hormonal therapy, targeted therapy, immunotherapy, or biological therapy).
  * Radiosurgery or radiotherapy. (Note: A tumor lesion situated in a previously irradiated area is considered a measureable/target lesion only if subsequent disease progression has been documented in the lesion.)
  * Initiation of a new erythropoietin, darbepoietin, and/or bisphosphonate therapy. (See Section 9.3.)
  * Minor surgery. (Note: Placement of a vascular access device is not considered minor or major surgery.)
  * Serious or uncontrolled infection.
  * Infection requiring parenteral antibiotics. (Note: Patients with a non-serious infection under active treatment and controlled with oral antibiotics initiated at least 10 days prior to initiation of protocol-indicated treatment are not excluded - e.g. urinary tract infection controlled with oral antibiotics.)
  * Unexplained fever > 38.0 ºC.
* ≤ 7 days before first dose of protocol-indicated treatment:

  * Receipt of granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF). (See Section 9.3.)
* Concurrent use of any medications or substances (e.g. herbal supplement or food) known to be a strong inhibitor or strong inducer of CYP3A4.

  * Although corticosteroids are considered to be strong inducers of CYP3A4, physiologic replacement doses of corticosteroids ≤ 10 mg daily prednisone or equivalent are allowed (Section 9).
* Inadequate recovery from toxicity attributed to prior anti-cancer therapy.

  * With the exception of alopecia, fatigue, or peripheral neuropathy, patients must have recovered to ≤ Grade 1 (NCI-CTCAE v5.0) residual toxicity prior to first dose of protocol-indicated treatment.
  * Patients requiring replacement therapy (e.g. prednisone or thyroid replacement therapy) for endocrine disorders from prior checkpoint inhibitor therapy are allowed
* Known history of allergy or intolerance which, in the opinion of the investigator, was an unacceptable adverse reaction attributed by the investigator to any prior anti-neoplastic therapy specifically targeting vascular endothelial growth factor or the VEGF receptor.
* Known history of allergy or intolerance which, in the opinion of the investigator, was an unacceptable adverse reaction attributed by the investigator to any prior anti-neoplastic therapy specifically targeting T-cell costimulation or immune checkpoint pathways - i.e. nivolumab (OPDIVO), pembrolizumab (KEYTRUDA), atezolizumab (TECENTRIQ), ipilimumab (YERVOY), etc.
* Non-healing wounds on any part of the body.
* Known or suspected clinically significant active bleeding.
* Inability to swallow oral medication; or the presence of a poorly controlled gastrointestinal disorder that could significantly affect the absorption of oral study drug - e.g. Crohn's disease, ulcerative colitis, chronic diarrhea (defined as > 4 loose stools per day), malabsorption, or bowel obstruction.
* patients with radiographic evidence of major airway or blood vessel invasion by cancer, radiographic evidence of intra-tumor cavitation, or gross hemoptysis (≥ one teaspoon) within the preceding 2 months.
* Significant cardiovascular disease or condition including:

  * Congestive heart failure (CHF) that is uncontrolled on current therapy.
  * Class III or IV cardiovascular disease according to the New York Heart Association (NYHA) Functional Criteria.
  * Uncontrolled arrhythmia.
  * Severe conduction disturbance (e.g. 3rd degree heart block).
  * Unstable angina pectoris (i.e. last episode ≤ 6 months prior to first dose of protocol-indicated treatment).
  * Uncontrolled (per investigator judgment) hypertension.
  * Myocardial infarction within 6 months prior to starting trial treatment.
  * QTcF >450 ms in men, or >470 ms in women.
* Deep vein thrombosis or pulmonary embolism ≤ 4 weeks before first dose of protocol-indicated treatment, unless adequately treated and stable.

  * Patients receiving therapeutic non-coumarin anticoagulation are eligible, provided they are on a stable dose (per investigator judgment) of anticoagulant.
* Patients with active interstitial lung disease and non-infectious pneumonitis or a history of active interstitial lung disease or pneumonitis requiring treatment with steroids or that may interfere with the detection or management of suspected drug-related pulmonary toxicity. Patients with lung cancer with a remote history (> 3 months ago) of pneumonitis following chemo-radiation treatment that has resolved are allowed.

Note: Patients with Chronic Obstructive Pulmonary Disease (COPD) whose disease is controlled (per investigator judgment) at trial entry are not excluded.

* CNS metastasis, unless asymptomatic and stable with no change in CNS disease status for at least two (2) weeks prior to initiating protocol-indicated treatment.

  * Anticonvulsant and/or corticosteroid prophylaxis (≤ 10 mg/day prednisone or equivalent daily) will be allowed if patient is on a stable or decreasing dose of such treatment for at least 14 days prior to initiating protocol-indicated treatment.
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone or equivalent daily) or other immunosuppressive medications within 14 days prior to initiating protocol-indicated treatment.

  * In the absence of active autoimmune disease: Subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhalational) ≤ 10 mg/day prednisone or equivalent daily; and physiologic replacement doses of systemic corticosteroids ≤ 10 mg/day prednisone or equivalent daily (e.g. hormone replacement therapy needed in patients with hypophysitis).
* Active, known or suspected autoimmune disease.

  * Subjects with type I diabetes mellitus; hypothyroidism; or endocrine disorders requiring hormone replacement even if due to prior immunotherapy; skin disorders such as vitiligo, psoriasis or alopecia not requiring systemic treatment; or conditions not expected by the investigator to recur in the absence of an external trigger are permitted to enroll.
* Uncontrolled (per investigator judgment) type I or type II diabetes mellitus.
* Known positive test for Human Immunodeficiency Virus (HIV) or known Acquired Immunodeficiency Syndrome (AIDS).
* Any active Hepatitis B or Hepatitis C infection.

  * Hepatitis B and C testing required ≤ 28 days prior to initiating protocol-indicated treatment, including at least: Hepatitis B surface antigen (HBV sAg); and Hepatitis C virus antibody (HCV Ab) or Hepatitis C virus RNA (HCV RNA).
* Solid tumor transplantation
* Immunization with any attenuated live vaccine within 1 week prior to initiating protocol-indicated treatment.
* Active second malignancy or history of a previous second malignancy within the last 2 years that could in the opinion of the investigator interfere with their assessment of study treatment.

  * Exceptions include the following permitted conditions - provided a complete remission was achieved at least 2 years prior to initiating protocol-indicated treatment AND no additional therapy (with the exception of allowable anti-estrogen/androgen therapy or bisphosphonates) is ongoing or required during the trial period: non-melanoma skin cancers (e.g. basal or squamous cell); superficial bladder cancer; or carcinoma in situ of the prostate, cervix, or breast.
* Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the investigator to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with and interpretation of scheduled visits, treatment schedule, laboratory tests and other study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Beckermann, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (7):
  - Stanford Cancer Institute, Palo Alto, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Escalation Level 1 (Vorolanib 200 mg +Nivolumab 240mg): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Vorolanib: Given by mouth
  Nivolumab: Given by IV
- Escalation Level 2 (Vorolanib 300mg + Nivolumab 240mg): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
- Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance: Participants receive 200mg vorolanib PO QD on days 1-56 and nivolumab 240mg IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Vorolanib: Given by mouth
  Nivolumab: Given by IV
- Dose Expansion - Non Small-Cell-Lung Cancer Naive; Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory; Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy; Dose Expansion - Thymic Carcinoma: Participants receive vorolanib 200mg PO QD on days 1-56 and nivolumab 240mg IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Vorolanib: Given by mouth
  Nivolumab: Given by IV
Period: Overall Study
Arm/Group | Escalation Level 1 (Vorolanib 200 mg +Nivolumab 240mg) | Escalation Level 2 (Vorolanib 300mg + Nivolumab 240mg) | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
Started | 3 | 7 | 19 | 15 | 17 | 18 | 9
Completed | 1 | 1 | 4 | 4 | 2 | 2 | 1
Not Completed | 2 | 6 | 15 | 11 | 15 | 16 | 8
Not completed — Death | 2 | 6 | 12 | 10 | 14 | 14 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Refused follow-up | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Declining Performance Status | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Still on study | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Undergoing radiation therapy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Escalation Level 1 (Vorolanib 200+Nivolumab 240mg): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Vorolanib: Given by mouth
  Nivolumab: Given by IV
- Escalation Level 2 (Vorolanib 300+Nivolumab 240mg): Participants receive vorolanib PO QD on days 1-56 and nivolumab IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
- Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance; Dose Expansion - Non Small-Cell-Lung Cancer Naive; Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory; Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy; Dose Expansion - Thymic Carcinoma: Participants receive vorolanib 200mg PO QD on days 1-56 and nivolumab 240mg IV over 30 minutes every two weeks (i.e. on Days 1, 15, 29, and 43 of each 56-day cycle) for the first two treatment cycles. After which, the treatment schedule can change to every four weeks (i.e., on Days 1 and 29 of each 56-day cycle) if the patient is not exhibiting disease progression.
  Vorolanib: Given by mouth
  Nivolumab: Given by IV
- Total: Total of all reporting groups
Arm/Group | Escalation Level 1 (Vorolanib 200+Nivolumab 240mg) | Escalation Level 2 (Vorolanib 300+Nivolumab 240mg) | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma | Total
Number analyzed (Participants) | 3 | 7 | 19 | 15 | 17 | 18 | 9 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 9 | 5 | 8 | 10 | 6 | 42
  >=65 years | 3 | 3 | 10 | 10 | 9 | 8 | 3 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 6 | 9 | 9 | 7 | 2 | 38
  Male | 3 | 2 | 13 | 6 | 8 | 11 | 7 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 3 | 7 | 16 | 15 | 12 | 16 | 8 | 77
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 5 | 2 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 4 | 1 | 2 | 1 | 9
  White | 3 | 7 | 17 | 10 | 13 | 15 | 5 | 70
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 19 | 15 | 17 | 18 | 9 | 88

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Combination Dose in Phase I (Per Common Terminology Criteria for Adverse Events (CTCAE) Criteria Version 5)
Description: Maximum tolerated dose for vorolanib daily combined with 240mg nivolumab every 2 weeks based on 3+3 dose escalation design. When 2 out of 6 patients at one dose experienced dose limiting toxicity, lower dose will be used.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: At 28 days
Population: 8 patients with NSCLC and 2 patients with TC who received vorolanib orally daily and 240mg nivolumab every 2 weeks, and had assessable results.
Measure: Number; unit: mg
Arm/Group | Escalation
Number analyzed (Participants) | 10
mg | 200

2. Primary Outcome: Objective Response Rate in Phase II.
Description: Antitumor activity will be assessed by objective response rate. Best response is determined as complete response(CR), partial response(PR), stable disease and progressive disease based on per Response Evaluation Criteria in Solid Tumors (RECIST). Objective response rate is the percentage of patients who had a CR or PR.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: Up to 1 year.
Population: Patients who received 200mg vorolanib daily with 240mg nivolumab every two weeks and were available for measurement of tumor response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
Number analyzed (Participants) | 18 | 15 | 17 | 18 | 9
percentage of participants | 11.1 [0 to 27.8] | 33 [13 to 60] | 5.9 [0 to 17.6] | 0 [0 to 0] | 11 [0 to 33]

3. Primary Outcome: Progression Free Survival in Phase II
Description: Antitumor activity will be assessed by progression free survival. Progression is termined per Response Evaluation Criteria in Solid Tumors (RECIST). Progression free survival (PFS) is defined as time from on treatment to disease progression or death (whicever comes first). Those without progression and alive were censored at last follow up. Kaplan-meier method is used to estimate the median survival time.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: Up to 1 year.
Population: Patients who received 200mg vorolanib daily with 240mg nivolumab every two weeks and were available for measurement of tumor response(progression).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
Number analyzed (Participants) | 18 | 15 | 17 | 18 | 9
months | 1.97 [1.54 to 4.60] | 7.16 [1.38 to NA] — insufficient number of participants with events | 3.22 [1.84 to 4.60] | 1.36 [0.92 to 1.81] | 9.1 [1.81 to NA] — insufficient number of participants with events

4. Primary Outcome: Duration of Response in Phase II.
Description: Duration of best response among patients who responsed to the treatment. Best response per Response Evaluation Criteria in Solid Tumors (RECIST). The duration of response was estimated from the first date of best overall response of a complete (CR) or partial response (PR) to the date of disease progression or death, using the Kaplan-Meier method.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: Up to 1 year
Population: Patients who received 200mg vorolanib daily with 240mg nivolumab every two weeks, were available for measurement of tumor response, and had partial or complete response. No patients in the "Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy" group had a partial or complete response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Thymic Carcinoma
Number analyzed (Participants) | 2 | 5 | 1 | 1
months | 2.7 [2.1 to NA] — Not enough patients and events for estimating. | NA [9.1 to NA] — Not enough events for estimating. | 12.8 [NA to NA] — Not enough patients and events for estimating. | NA [NA to NA] — Not enough patients and events for estimating.

5. Primary Outcome: Disease Control Rate in Phase II. Best Response Per Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Antitumor activity will be assessed by disease control rate. Best response (complete response,CR; partial response, PR;stable disease , SD; or progression,PD) per Response Evaluation Criteria in Solid Tumors (RECIST). Disease control rate is the percentage of patients who had a CR,PR or SD.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: Up to 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
Number analyzed (Participants) | 18 | 15 | 17 | 18 | 9
percentage of participants | 44.4 [22.2 to 66.7] | 53.3 [26.7 to 80.0] | 52.9 [29.4 to 76.5] | 11.0 [0 to 27.8] | 66.7 [33.3 to 100]

6. Primary Outcome: Overall Survival in Phase II.
Description: Antitumor activity will be assessed by overall survival. Overall survial is defined as the time from on treatment to death. Those alive were censored at last follow up. Kaplan-meier method is used to estimate the median overall survival time.
  We have specified the phase I and phase II populations as study arms; note outcome measures are then distinct for each arm, with the phase I arm intended to assess safety (MTD), and the phase 2 arm intended to assess efficacy, as typical for phase I-II studies. Thus, for each outcome, only the phase I cohort is included in the analysis population, or only the phase II cohort is including in the analysis population, as relevant to the outcome measure.
Time Frame: Up to 2 years.
Population: Patients who received 200mg vorolanib daily with 240mg nivolumab every two weeks and were available for measurement of survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
Number analyzed (Participants) | 18 | 15 | 17 | 18 | 9
months | 10.81 [4.60 to NA] — insufficient number of participants with events | NA [8.77 to NA] — insufficient number of participants with events | 16.27 [5.98 to NA] — insufficient number of participants with events | 4.5 [3.75 to NA] — insufficient number of participants with events | 21.06 [13.54 to NA] — insufficient number of participants with events

7. Other Pre Specified Outcome: Correlation Between Biomarkers and Response for Phase II Patients
Description: Antitumor activity will be assessed by correlation between the biomarkers and clinical outcomes. This is a exploratory end point. To assess the effects of combinatorial treatment on specific pharmacodynamic and pharmacogenetic biomarkers, including but not limited to circulating levels of serum CSF1 and VEGF, protein expression using CyTOF, and multiplex immunofluorescence.
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initiation of protocol-indicated treatment up to approximately 67 months.
Arm/Group | Escalation Level 1 (Vorolanib 200+Nivolumab 240mg) | Escalation Level 2 (Vorolanib 300+Nivolumab 240mg) | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance | Dose Expansion - Non Small-Cell-Lung Cancer Naive | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy | Dose Expansion - Thymic Carcinoma
All-Cause Mortality (participants affected / at risk) | 2/3 | 6/7 | 13/19 | 12/15 | 14/17 | 14/18 | 4/9
Serious Adverse Events (participants affected / at risk) | 3/3 | 6/7 | 9/19 | 10/15 | 9/17 | 5/18 | 6/9
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 19/19 | 15/15 | 17/17 | 18/18 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Level 1 (Vorolanib 200+Nivolumab 240mg) (N=3) | Escalation Level 2 (Vorolanib 300+Nivolumab 240mg) (N=7) | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance (N=19) | Dose Expansion - Non Small-Cell-Lung Cancer Naive (N=15) | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory (N=17) | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy (N=18) | Dose Expansion - Thymic Carcinoma (N=9)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 2 (2) | 3 (5) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epidural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Port infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered mental state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic volume overload (administration site) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thymic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (3) | 0 (0) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volume depletion (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hip pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurex catheter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Pericardial Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Exacerbation of COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fractured ankle (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus of Gallbladder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chronic Venous Stasis ulcer (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurx catheter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral hepatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracoscopy Pericaridal window (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation Level 1 (Vorolanib 200+Nivolumab 240mg) (N=3) | Escalation Level 2 (Vorolanib 300+Nivolumab 240mg) (N=7) | Dose Expansion - Non Small-Cell-Lung Cancer Acquired Resistance (N=19) | Dose Expansion - Non Small-Cell-Lung Cancer Naive (N=15) | Dose Expansion - Non Small-Cell-Lung Cancer Primary Refractory (N=17) | Dose Expansion - Small Cell Lung Cancer - Progressed on Platinum-based Chemotherapy (N=18) | Dose Expansion - Thymic Carcinoma (N=9)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 1 (2) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3) | 0 (0) | 4 (5) | 2 (4) | 1 (1) | 4 (4)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (4) | 5 (6) | 11 (12) | 5 (8) | 8 (12) | 9 (9) | 3 (6)
Limb edema (General disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (5) | 1 (3) | 2 (2) | 2 (2)
Fever (General disorders) | 2 (6) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Pulminary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (5) | 7 (8) | 2 (3) | 1 (1) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pleura effustion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound on left heel post surgery (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tripped (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Possible spider bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular fungal infection (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 2 (3) | 0 (0) | 3 (3)
Seasonal allegies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 1 (3)
Hypertenson (Vascular disorders) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 3 (3) | 2 (3) | 2 (4)
Hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Virus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (7) | 4 (5) | 4 (4) | 0 (0) | 1 (1)
Sclerosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (20) | 3 (5) | 2 (3) | 5 (7)
Constrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 5 (6) | 7 (17) | 5 (8) | 3 (3) | 2 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (8) | 5 (5) | 4 (9) | 8 (10) | 3 (3) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (8) | 1 (3) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Face edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 3 (6) | 6 (12) | 2 (7) | 1 (2) | 5 (18)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (6) | 2 (4) | 6 (14) | 3 (7) | 3 (4) | 7 (19)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (3) | 0 (0) | 1 (1) | 4 (6)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Urine leukocyte esterase (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sacral lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae on fingers and chest (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 11 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (7) | 1 (1) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 4 (14) | 2 (12) | 2 (7) | 0 (0) | 1 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 2 (11) | 3 (4) | 1 (1) | 1 (3)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (8) | 2 (2) | 2 (2) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 3 (10) | 2 (16) | 3 (15) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 0 (0) | 2 (2) | 0 (0)
Elevated LFTs (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Esophogeal stricture (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peeling finger tips (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair color change (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left hip total arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected root canal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aches in legs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aches in neck (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vaginal yeast (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left shoulder nodule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Blood bilirubin increased (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated AST and ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transaminitis (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Glucose intolerence (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Tremor in left hand (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningismus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Left mid-back skin nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash on back of head (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small red pinpoint rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Yeast under both breasts (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Itching under both breasts (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial wound on left back of calf (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulled right big toe nail off (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pacemaker placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Port-a-cath placed in rt. internal jugular (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testosterone deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular migrane (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Klebsilla Pneumoniae (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased sodium (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated bilirubin (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restlessness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated TSH (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Stool color change (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach flu (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loose stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trunk edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Umbilical Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Common cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic toxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection of the hypopharynx and larynx (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Right hand cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left side rib pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Falling backward sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilateral Hand Numbness/Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head cold (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itchy throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash, left buttocks (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
R supraclavicular fullness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary vasospasm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03583086/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT03583086/ICF_000.pdf